CLINICAL TRIAL: NCT05327777
Title: Toward Zero Prescribed Opioids for Outpatient General Surgery Procedures: a Prospective Cohort Trial
Brief Title: Toward Zero Prescribed Opioids for Outpatient General Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19D.688
Record Dates: First submitted 2022-04-01; First posted 2022-04-14 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Opioid Misuse and Addiction; Pain
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Pain | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Control group, opioid sparing arm, and zero opioid arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Normal standard practices
- Opioid Sparing (Experimental): Providers required to prescribe 10 narcotic pills only
  Interventions: Drug: Oxycodone
- Zero Opioid (Experimental): No narcotic prescription is provided to patient at discharge
  Interventions: Behavioral: Zero Opioid Protocol

INTERVENTIONS:
Drug: Oxycodone — Investigators provided set opioid prescriptions for 10 pills each patient.
  Arms: Opioid Sparing
Behavioral: Zero Opioid Protocol — Investigators provided no opioid prescriptions at discharge and instead provided information on non-narcotic pain control.
  Arms: Zero Opioid

SUMMARY:
Investigators have created an opioid reduction "package" which includes patient education, non-narcotic pain control instructions, and limited (or no) opioid pain prescriptions provided at discharge in an attempt to reduce the number of opioid consumption after outpatient general surgery.

DETAILED DESCRIPTION:
Between November 2019 and July 2021, patients undergoing elective inguinal hernia repair (IHR) or cholecystectomy were enrolled in the study. Patients were divided into three cohorts: Control, opioid sparing (OS), or zero-opioid (ZO). Control patients did not have any intervention; OS patients had an opioid reduction intervention protocol applied (patient education and perioperative multimodal analgesia) and were provided an opioid prescription at discharge; the ZO had the same protocol, however patients were not provided opioid prescriptions at discharge. Two weeks after discharge patients were interviewed to record opioid consumption, pain scores, and level of satisfaction since discharge.

ELIGIBILITY:
Inclusion Criteria:

* Opioid naïve patients
* Age > 18
* Being scheduled for an outpatient elective inguinal hernia repair or cholecystectomy

Exclusion Criteria:

* Urgent/emergent status
* Previous cholecystostomy tube placement

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Palazzo, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No Plans to share the IPD

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Opioid Sparing | Zero Opioid
Started | 58 | 42 | 29
Completed | 58 | 42 | 29
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Opioid Sparing | Zero Opioid | Total
Number analyzed (Participants) | 58 | 42 | 29 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (1.8) | 55.3 (2.0) | 58.6 (2.9) | 54 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 2 | 31
  Male | 39 | 32 | 27 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 7 | 15
  White | 47 | 31 | 22 | 100
  More than one race | 5 | 4 | 0 | 9
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 58 | 42 | 29 | 129
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 27.8 [25.4 to 32.1] | 27.9 [24.3 to 31] | 25.4 [23.3 to 28.7] | 27 [25 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Morphine Milligram Equivalents Taken by Participants
Description: Patients will be interviewed fourteen days after procedure and asked how many opioid pills they have taken since being discharged form the hospitals
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Control | Opioid Sparing | Zero Opioid
Number analyzed (Participants) | 58 | 42 | 29
morphine milligram equivalents | 46 [37.5 to 75] | 15 [11 to 22.5] | 0 [0 to 0]

2. Secondary Outcome: Satisfaction Scores Ranging From 1 - 10
Description: Patient will be asked to rank their satisfaction scores on a scale from 1 - 10 (with 1 being extremely dissatisfied and 10 being extremely satisfied) since discharge from the hospital
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | Opioid Sparing | Zero Opioid
Number analyzed (Participants) | 58 | 42 | 29
units on a scale | 10 [9 to 10] | 10 [9 to 10] | 10 [8.5 to 10]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Does not differ
Arm/Group | Control | Opioid Sparing | Zero Opioid
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/42 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/42 | 0/29
Other Adverse Events (participants affected / at risk) | 0/58 | 0/42 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT05327777/Prot_SAP_004.pdf